CLINICAL TRIAL: NCT02895542
Title: Preparatory Work to Assess Adherence to Oral Chemotherapy Among Patients With Chronic Myeloid Leukemia
Brief Title: Preparatory Work to Assess Adherence to Oral Chemotherapy
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00039112; REBAWF 99716CD (Other: NCI)
Record Dates: First submitted 2016-09-06; First posted 2016-09-09 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oral Anti-Cancer Agent: No intervention

SUMMARY:
This study to find out more about how patients take their anticancer medications and challenges related to taking cancer medications.

DETAILED DESCRIPTION:
120 patients with Chronic Myeloid Leukemia (CML) who are currently prescribed an oral anti-cancer agent from up to 6 CCDR NCORP sites to complete a brief interviewer administered survey to assess medication adherence and related factors.

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed with Chronic Myeloid Leukemia (CML) and is receiving care for CML at a participating CCDR NCORP practice,
* Patient had been prescribed one of the following oral anticancer agents for CML for ≥30 days (Imatinib, Nilotinib, Dasatinib, Bosutinib, Ponatinib). Prior use of any of these medications is allowed, as long as they have been on a stable regimen for at least 30 days prior to enrollment.
* Patient is 18 years of age or older

Exclusion Criteria:

* Patient does not speak English or requires an interpreter for medical visits
* Patient is cognitively impaired, as determined by the referring provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Conducting brief structured interviews, to further understand potential patient characteristics and barriers associated with non-adherence of medication. With this knowledge of identified patient barriers, interventional strategies can be designed to improve CML care, monitoring and adherence.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Patient Demographic and Health Behaviors Questionnaire | Study 1 day Visit
  Questions will be asked about the participants demographic background and health behaviors.
Brief Medication Questionnaire (BMQ) | Study 1 day Visit
  A self-report tool for screening adherence and barriers to adherence. The tool includes a 5-item Regimen Screen that asks patients how they took each medication in the past week, a 2-item Belief Screen that asks about drug effects and bothersome features, and a 2-item Recall Screen about potential difficulties remembering.
Single Item Adherence Measure 1 | Study 1 day Visit
  This is a single question. This measure was developed to serve as simple means of identifying sub-optimal adherence which could help identify at-risk patients for interventions.
Single Item Adherence Measure 2 | Study 1 day Visit
  This single item was developed to evaluate self-report adherence to medication and has demonstrated low patient burden and the ability to predict adherence-related clinical outcomes as good or better than other adherence measures.

SECONDARY OUTCOMES:
REALM-SF | Study 1 day Visit
  The REALM-SF offers researchers a simplified, validated, and efficient instrument for assessing patient literacy in clinical setting. It can be used to investigate the relationship between literacy and specific health outcomes such as medication adherence and health care utilization.
Medications Adherence Reasons Scale (MARS) | Study 1 day Visit
  This questionnaire is designed to identify potential risk factors associated with medication-related non-adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Weaver, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No